CLINICAL TRIAL: NCT02560909
Title: A Randomized Controlled Trial Comparing Adjuvanted vs. Nonadjuvanted Influenza Vaccine in Adult Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Recipients.
Brief Title: Adjuvanted Influenza Vaccine in Stem Cell Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Physician, Transplant Infectious Diseases, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-9503
Record Dates: First submitted 2015-09-03; First posted 2015-09-25 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Transplantation; Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will receive one dose MF59 adjuvanted intramuscular vaccine.
  Interventions: Biological: FLUAD® influenza vaccine
- Control (Active Comparator): The control group will receive one dose of the standard 2015-2016 nonadjuvanted vaccine.
  Interventions: Biological: FLUVIRAL®

INTERVENTIONS:
Biological: FLUAD® influenza vaccine — MF59 adjuvant has been used in seasonal influenza vaccine in Canada and Europe for people ≥65 years. MF59 contains squalene, polysorbate 80, and sorbitan trioleate. It is packaged as small microvesicles of 160nm diameter. The complete mechanism of action of MF59 is not well understood but requires activation of the innate immune system; the adjuvant exerts a local inflammatory response increasing the influx of neutrophils and macrophages to the injection site.
  Other Names: MF59 adjuvanted vaccine
  Arms: Experimental
Biological: FLUVIRAL® — Standard 2015-2016 nonadjuvanted vaccine
  Other Names: Trivalent Influenza Vaccine
  Arms: Control

SUMMARY:
Influenza virus is an important cause of morbidity in the transplant population and can lead to viral and bacterial pneumonia. Although the annual influenza vaccine is recommended for transplant patients, studies have shown that nonadjuvanted vaccine has poor immunogenicity. There are no studies that define the effect of adjuvanted vaccine in this population. The purpose of this study is to determine if a vaccination with FLUAD® results in improved immunogenicity as compared to standard vaccine in allo-HSCT recipients. Immunogenicity will be assessed by standard quantitative antibody titer assessments and using cell-mediated immunity measurements.

DETAILED DESCRIPTION:
The investigators plan to study the immunogenicity of two different types of the influenza vaccine in 240 allogeneic stem cell transplant patients during the 2015-2016 season. Patients will be randomized to receive either adjuvanted influenza vaccine or nonadjuvanted. Antibody titers will be evaluated by a standard hemagglutination inhibition assay. The investigators hypothesize that the patients who receive the adjuvanted influenza vaccine will reach significantly higher response to the vaccine. This study advances research on the prevention of serious viral infections in transplant recipients.

Results from this study have the potential to directly improve patient care. If the use of the adjuvanted influenza vaccine is successful, this strategy may lead to a significant reduction in burden of disease, hospitalizations, and long-term morbidity.

The co-administration of vaccine with an adjuvant is a potentially promising method of boosting immunogenicity. Two adjuvants have been used in influenza vaccines: AS03 and MF59. Both are oil-in-water emulsions. AS03 was used in the monovalent pandemic A/H1N1 vaccine in Canada and Europe. Adjuvanted vaccines have been studied in the hematopoietic stem cell transplant population with most studies done in using the AS03-adjuvanted pandemic vaccine. MF59 adjuvant has been used in seasonal influenza vaccine in Canada and Europe for people ≥65 years old. MF59-adjuvanted vaccines have not been well studied in hematopoietic stem cell transplantation but could represent a significant advance if they show greater immunogenicity than the standard non-adjuvanted influenza vaccine. Both FLUAD® and the standard 2015-2016 nonadjuvanted vaccine will contain 15 microgram antigen from each strain and will be injected in a standard dose (0.5 mL) in the deltoid muscle by trained personnel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Greater than 3 months post-transplant
* Allogeneic HSCT

Exclusion Criteria:

* Has already received influenza vaccination for 2015-2016 season
* Egg allergy
* Previous life-threatening reaction to influenza vaccine (i.e. Guillain Barre Syndrome)
* Febrile illness in the past one week
* Receipt of intravenous immunoglobulin (IVIG) in the past 30 days or planning to receive IVIG in the next 4 weeks
* Unable to provide informed consent
* Unable to comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rates of seroconversion | 4 weeks from vaccination
  serological response with a four-fold or greater increase in HI antibody titers to an antigen

SECONDARY OUTCOMES:
Rates of seroprotection | 4 weeks from vaccination
  HIA titers of >=1:40
Rate of Local and systemic adverse events to vaccination | within 7 days of vaccination
Number of participants with microbiologically-documented influenza infection | 6 months from vaccination
  confirmed by direct fluorescent antibody, viral culture, or PCR

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No